CLINICAL TRIAL: NCT03674515
Title: Study of Program Interest "Bouge" to Improve the Daily Physical Activity and Tolerance in Processings Treatment of Non-metastatic Breast Cancer at the Beginning Weekly Taxol Adjuvant Chemotherapy (Www.Bouge-coaching.Com)
Brief Title: Study of Program Interest "Bouge" to Improve the Daily Physical Activity in Processings Treatment of Non-metastatic Breast Cancer
Acronym: BOUGE CANCER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BOUGE CANCER (29BRC17.0038)
Record Dates: First submitted 2018-02-19; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Physical Activity; Breast Cancer; Mobile Health Apps
MeSH Terms: conditions — Motor Activity; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Smartphone application "placebo"
  Interventions: Device: Smartphone application "placebo"
- "Bouge" (Active Comparator): Smartphone equipped with the application "Bouge"
  Interventions: Device: Smartphone equipped with application "bouge" = Coach group

INTERVENTIONS:
Device: Smartphone application "placebo" — Strategy based on smartphone application "placebo"
  Arms: placebo
Device: Smartphone equipped with application "bouge" = Coach group — Strategy based on smartphone application "bouge"
  Arms: "Bouge"

SUMMARY:
Evaluate the "Bouge" digital program (smartphone application) to increase the daily physical activity of breast cancer patients

DETAILED DESCRIPTION:
Controlled, randomized, open, prospective, multicentric study, 214 volunteer patients aged between 18 and 70, with breast cancer, at the start of TAXOL treatment, possessing a smartphone, will be recruited and randomized into two groups:

107 in the control group (smartphone application "placebo" = number of steps) 107 will be equipped with the application "Bouge" = coached group

For three months, the patients do their daily physical activity. The "coached" group, through the smartphone application "Bouge", receives computer coaching to increase their physical activity (no direct medical intervention, only notifications and computer pusch).

The control group is not coached by the application (simple display of the number of step)

ELIGIBILITY:
Inclusion Criteria:

non-metastatic breast cancer start of treatment with TAXOL compatible smartphone

Exclusion Criteria:

age metastatic breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-12 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Increased daily physical activity (number of steps) using the smartphone application "BOUGE" | 12 weeks
  The objective is an increase of 3000 steps daily between J 1 and J 90 (an increase of 15 000 steps between S1 and S 12)

SECONDARY OUTCOMES:
Well-being, | 12 weeks
  Scale EQ-5D-5L,
Well-being, | 12 weeks
  Scale EORTC QLQ-C30,
Fatigue | 12 weeks
  Scale WHO
Sleep | 12 weeks
  Scale SPIEGEL

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CHU de Morlaix, Morlaix